CLINICAL TRIAL: NCT07209800
Title: Effectiveness of Whole-Body Sensory Integration Therapy on Chewing Function and Feeding Behaviors in Children With Chewing Disorders
Brief Title: Sensory Therapy for Chewing in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Neslihan Altuntas Yilmaz, Assistant Professor, PhD, Necmettin Erbakan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEU-PT2025-01
Record Dates: First submitted 2025-09-29; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Chewing Difficulties in Children; Feeding Behavior Challenges; Oral-motor Dysfunction; Impaired Chewing Function
Keywords: Chewing disorder, Karaduman Chewing Performance Scale (KCPS), Oral awareness, Pediatric rehabilitation, Sensory integration therapy.

STUDY DESIGN:
Intervention Model Description: This study was conducted as an experimental, single-group, pretest-posttest design. Participants received whole-body sensory integration therapy, and pre- and post-intervention assessments were used to evaluate changes in chewing function and feeding behaviors
Masking Description: The outcomes assessor was blinded; the researcher administering the intervention was not involved in the assessments
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sensory integration therapy (Experimental): Sensory integration therapy (SIT) was delivered individually in a play-based format, three times per week for four weeks, totaling 12 sessions. Each session lasted 60 minutes, and parents were instructed to reinforce the activities at home as homework. All interventions were administered one-on-one by an experienced therapist in a therapy room. The therapist who administered the intervention did not take part in the evaluation process; therefore, the study was conducted in a single-blind manner. Before the intervention, a trust-based relationship was established with the children, and sensory activities were performed within a play context. The interventions were not limited to oral activities but aimed to support overall sensory development [8]. Based on this program, sensory integration procedures were applied at regular intervals.
  Interventions: Other: Sensory integration therapy

INTERVENTIONS:
Other: Sensory integration therapy — Sensory integration therapy (SIT) was delivered individually in a play-based format, three times per week for four weeks, totaling 12 sessions. Each session lasted 60 minutes, and parents were instructed to reinforce the activities at home as homework. All interventions were administered one-on-one by an experienced therapist in a therapy room. The therapist who administered the intervention did not take part in the evaluation process; therefore, the study was conducted in a single-blind manner. Before the intervention, a trust-based relationship was established with the children, and sensory activities were performed within a play context. The interventions were not limited to oral activities but aimed to support overall sensory development [8]. Based on this program, sensory integration procedures were applied at regular intervals.

SUMMARY:
Brief Summary

The goal of this study is to learn if whole-body sensory integration therapy can improve chewing skills and mealtime behaviors in children with chewing difficulties. The main questions it aims to answer are:

Does the therapy help children chew food better?

Does it make mealtimes shorter and more efficient?

Participants will:

Attend individual sensory integration therapy sessions for 60 minutes, three times a week for 4 weeks

Take part in exercises such as vibration, crawling through a tunnel, therapeutic brushing, joint and oral exercises, and sensory activities

Be observed for chewing performance and report meal duration and daily meal frequency before and after the therapy

Researchers will compare the results from before and after the therapy to see if chewing skills and feeding behaviors improve.

DETAILED DESCRIPTION:
Detailed Description

The aim of this study is to evaluate the effectiveness of whole-body sensory integration therapy on chewing function, meal duration, and feeding behaviors in children with chewing difficulties. Chewing difficulties in children can arise from developmental disorders, such as cerebral palsy, autism spectrum disorder, or other neuromotor impairments. These difficulties can negatively affect nutritional intake, growth, and overall quality of life.

This study will include 31 children aged between 3 and 12 years who exhibit observable challenges in chewing or feeding. Participants will be randomly assigned to either an intervention group or a control group. The intervention group will receive whole-body sensory integration therapy three times per week for 4 weeks. Each therapy session will last approximately 60 minutes and include activities designed to enhance oral-motor function, chewing skills, body coordination, balance, and sensory processing. Examples of therapy activities include:

Chewing exercises using therapy tools (e.g., chewing sticks, textured foods)

Oral-motor exercises to strengthen lips, tongue, and jaw muscles

Proprioceptive and vestibular activities such as crawling, climbing, balancing, and swinging

Play-based tasks that integrate sensory input with functional feeding activities

Parents or caregivers will be guided to support therapy exercises at home to reinforce skill acquisition.

Outcome measures will be collected at baseline and after the 4-week intervention. The primary outcome is improvement in chewing function, assessed using standardized tools suitable for pediatric populations. Secondary outcomes include changes in meal duration, frequency of meals, and overall feeding behaviors.

It is hypothesized that children receiving whole-body sensory integration therapy will demonstrate significant improvements in chewing efficiency, reduced meal times, and enhanced feeding behaviors compared to the control group. This study aims to provide evidence for the inclusion of sensory integration therapy as a clinical intervention to support feeding skills in children with chewing difficulties.

ELIGIBILITY:
Inclusion Criteria:

* Children with chewing difficulties aged around 5 years (approx. 55-69 months, based on mean ± SD)
* Medically stable and able to participate in feeding sessions
* Parental consent obtained

Exclusion Criteria:

* Children with severe medical conditions or genetic syndromes affecting feeding
* Children receiving other intensive feeding or sensory interventions during the study
* Inability to sit or participate in the evaluation sessions

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Chewing performance: | Pre-intervention assessment: Before the start of the therapy. Post-intervention assessment: Immediately after the completion of the therapy program (4 weeks).
  Assessed using the Karaduman Chewing Performance Scale (KCPS).
Meal frequency and duration | Pre-intervention assessment: Before the start of the therapy. Post-intervention assessment: Immediately after the completion of the therapy program (4 weeks).
  Average daily meal frequency and meal duration recorded via parent interviews.
Sociodemographic data: | Before the start of the therapy.
  Age, sex, height, weight, and diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Neslihan Altuntaş Yılmaz, Assistant Professor, Principal Investigator — Necmettin Erbakan University; Ahmet Sami Güven, Professor, Study Director — Necmettin Erbakan University
Locations (1):
- Nezahat Keleşoğlu Faculty of Health Sciences, Konya, Meram, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The study is complete; however, individual participant data (IPD) will not be publicly shared to protect participant confidentiality and ensure the security of personal data. Ethical approvals and consent forms do not cover data sharing. If requested, the corresponding author may share data on a case-by-case basis, ensuring participant confidentialit